CLINICAL TRIAL: NCT00246662
Title: Phase 1b Open-Label, Multicenter Clinical Study of the Safety and Activity of Intravenous Administration of SNS-595 in Patients With Advanced Hematologic Malignancies
Brief Title: Safety Assessment of Two Schedules of Intravenous Infusions of SNS-595 for the Treatment of Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunesis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPO-0004
Record Dates: First submitted 2005-06-30; First posted 2005-10-31 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Leukemia, Lymphocytic, Acute; Leukemia, Nonlymphocytic, Acute; Leukemia, Myeloid, Chronic; Myelodysplastic Syndromes
Keywords: Leukemia; Hematologic; Blood; Cancer; Malignancy; Myelodysplastic Syndromes
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Leukemia; Neoplasms | interventions — vosaroxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sch A (18 mg/m2 vosaroxin initially) (Experimental): Once weekly intravenous on days 1, 8, 15 up to 4 cycles
  Interventions: Drug: Vosaroxin
- Sch B (9 mg/m2 vosaroxin initially) (Experimental): Twice weekly intravenous administration on days 1, 4, 8, 11 up to 4 cycles
  Interventions: Drug: Vosaroxin

INTERVENTIONS:
Drug: Vosaroxin — All patients receive vosaroxin Injection
  Other Names: SNS-595; Voreloxin

SUMMARY:
This study primarily determined the safety and tolerability of escalating doses of vosaroxin (SNS-595) in 2 dose schedules, and assessed the PK profile of vosaroxin and defined a recommended dose regimen for Phase 2 studies. Secondarily the study assessed potential biomarkers and antileukemic activity.

DETAILED DESCRIPTION:
Patients assigned to 1 of 2 schedules (A and B) in cohorts of at least 3 patients received vosaroxin (SNS-595) intravenously (IV) for up to 4 cycles: once weekly (Days 1, 8, 15 in Schedule A) or twice weekly (Days 1, 4, 8, 11 in Schedule B). Dose escalation proceeded independently for Schedule A (18 mg/m2 initially) and Schedule B (9 mg/m2 initially) in the absence of Dose-limiting Toxicity (DLT) based on a modified Fibonacci sequence. The incidence of DLT during Cycle 1 determined the maximum-tolerated dose (MTD) allowing for treatment delays of up to 14 days to resolve clinically significant abnormal laboratory values or related treatment-emergent adverse events (TEAEs) and one dose reduction of 25% in case of above. Patients with stable disease, hematologic improvement, or partial remission with stable blast counts or experiencing clinical benefit in the opinion of the investigator were eligible to receive vosaroxin for up to 4 additional cycles.

ELIGIBILITY:
Inclusion:

* Able to understand and willing to sign a written informed consent document
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1, 0r 2
* Received less than or equal to 3 induction/re-induction regimens for disease(s) defined by the protocol
* Must have relapsed or refractory leukemia for which no standard therapies are expected to result in a durable remission; patients who have not received prior treatment who have either refused or, in the opinion of the Investigator, are not able to tolerate, standard therapy may be included.

Exclusion:

* Prior exposure to SNS-595 (vosaroxin)
* Pregnant or breastfeeding
* Women of childbearing potential or male partners of women of childbearing potential unwilling to use an approved, effective means of contraception according to the institution's standards
* Any evidence of active central nervous system (CNS) leukemia
* Any evidence of acute or chronic graft-versus-host disease
* Has active cancer (other than that which is defined by the inclusion criteria for this protocol), except for skin cancer (excluding melanoma)
* Laboratory values outside normal or reasonable reference range specified by the protocol
* Liver function and kidney function outside limits specified by the protocol
* Not yet recovered from side effects of previous cancer therapy
* Myocardial infarction, cerebrovascular accident/transient ischemic attack (TIA) or thromboembolic event (deep vein thrombosis or pulmonary embolus) within 6 months before the first SNS-595 dose
* Requires kidney dialysis (hemodialysis or peritoneal)
* Received an investigational agent within 14 days before Cycle 1, Day 1
* Prior pelvic radiation therapy or radiation to greater than or equal to 25% of bone marrow reserve (palliative radiation is not excluded as long as it does not exceed greater than or equal to 25% of bone marrow reserve)
* Any other medical (uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia), psychological, or social condition that, in the opinion of the Principal Investigator, would contraindicate the patient's participation in the clinical trial due to safety or compliance with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2005-11-14; Primary Completion 2008-12-23 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 6 months

SECONDARY OUTCOMES:
Pharmacokinetic profile | 6 months
Duration of leukemia-free survival | 6 months
Anti-tumor activity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Michelson, MD, Study Director — Sunesis Pharmaceuticals
Locations (5):
- United States (5):
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - University of Texas, MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Aggregate data of participants experiencing Adverse Events